CLINICAL TRIAL: NCT05345223
Title: A Registry Study on Primary/idiopathic Triglyceride Deposit Cardiomyovasculopathy
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Osaka University Graduate School of Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20334(T2)-3
Record Dates: First submitted 2022-03-29; First posted 2022-04-25 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Triglyceride Deposit Cardiomyovasculopathy
Keywords: triglyceride deposit cardiomyovasculopathy; TGCV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TGCV: Patients who have been confirmed as TGCV by a cardiologist.

SUMMARY:
The objective of this study is to construct a registry; in order to understand the onset status of triglyceride deposit cardiomyovasculopathy (TGCV) in Japan with patients' background and natural history of the disease, and to explore disease-specific prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have been conﬁrmed as TGCV based on the diagnostic criteria for TGCV

Exclusion Criteria:

* The patients who refused to participate in the study by opt-out

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (excluding under 20 years old) who have been confirmed as TGCV based on the diagnostic criteria for TGCV by a cardiologist.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The period between the date of TGCV diagnosis and the date of death due to any cause | 10 years
  The period is from the date of diagnosis of TGCV to the date of death due to any cause. Survival and lost follow-up cases will be censored on the final confirmation date of survival.

SECONDARY OUTCOMES:
Comparison of subjective symptoms, laboratory findings, and event occurrence before and after tricaprin therapy: Washout rate of BMIPP (%) | 10 years
Comparison of subjective symptoms, laboratory findings, and event occurrence before and after tricaprin therapy: LVEF (%) (UCG or QGS) | 10 years
Comparison of subjective symptoms, laboratory findings, and event occurrence before and after tricaprin therapy: Any cardiovascular events | 10 years
Presence (date of occurrence or treatment) or absence of various events | 10 years
  To measure the period from the date of diagnosis of TGCV to the date the following event occurs: non-fatal myocardial infarction by the outcome assessment, non-fatal stroke, hospitalization for heart failure, CABG, PCI, TVR, pacemaker/ICD implantation, CRT, VAD, acute coronary syndrome requiring hospitalization, hospitalization/device activation/heart transplantation due to fatal arrhythmia. However, surgery scheduled at the time of diagnosis will not be treated as an event.

CONTACTS AND LOCATIONS:
Overall Officials: Ken-ichi Hirano, MD, PhD, Principal Investigator — Department of Triglyceride Science, Graduate School of Medicine, Osaka University
Locations (7):
- Japan (7):
  - Aichi Medical University, Nagakute, Aichi-ken
  - Nagoya University, Nagoya, Aichi-ken
  - Chiba University Graduate School of Medicine, Chiba, Chiba
  - Kyushu University, Fukuoka, Fukuoka
  - Hyogo Medical University, Nishinomiya, Hyōgo
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University, Bunkyo, Tokyo